CLINICAL TRIAL: NCT01936194
Title: The Effects of Polyunsaturated Fatty Acids on Allergic/Atopic Dermatitis
Brief Title: The Effects of Polyunsaturated Fatty Acids (PUFA) on Allergic/Atopic Dermatitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators don't want to conduct this study as time is limited.
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: International Peace Maternity and Child Health Hospital (Other); Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 6018
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Docosahexaenoic Acid (DHA) (Experimental): infants receiving capsule containing DHA.
  Interventions: Dietary Supplement: DHA
- High Olive Oil (Other): infants receiving capsule without DHA and EPA.
  Interventions: Dietary Supplement: High Olive Oil
- DHA+EPA (Experimental): infants receiving capsule containing DHA and EPA.
  Interventions: Dietary Supplement: DHA+EPA

INTERVENTIONS:
Dietary Supplement: DHA+EPA
  Arms: DHA+EPA
Dietary Supplement: High Olive Oil
  Arms: High Olive Oil
Dietary Supplement: DHA
  Arms: Docosahexaenoic Acid (DHA)

SUMMARY:
This clinical trial will study the effects of PUFA supplementation during pregnancy and lactation period on fatty acid composition in human milk and plasma of the mothers and the clinical outcome of atopic dermatitis in infants at increased risk.

ELIGIBILITY:
Inclusion Criteria:

* Woman is pregnant between 16 and 20 weeks
* Mother delivers after 36 weeks
* Mother is willing to breast-feed for four months
* Mother has potential to deliver a child with increased risk of atopic dermatitis
* Signed Informed Consent

Exclusion Criteria:

* Mother is smoking
* Disease with influence on breast feeding
* Complicated pregnancy
* Allergic to seafood
* Allergic to soy
* Allergic to marine fish
* Mother has more than two salmon or tuna meals per week
* Mother is undergoing treatment with anticoagulants

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Lipid Analysis | Baseline, Delivery, Within one week after delivery, 6 weeks postpartum, 4 months postpartum
Metabolomics Study of PUFA | Baseline, Delivery, Within one week after delivery, 6 weeks postpartum, 4 months postpartum, 12 months postpartum
Skin Prick Test to Common Allergens | 4 months postpartum, 12 months postpartum
Clinical Assessment of IgE-mediated Allergic Eczema | 4 months postpartum, 12 months postpartum

SECONDARY OUTCOMES:
Fatty Acid Desaturase (FADS) Genotypes | Baseline
immunoglobulin E immunoglobulin E Immunoglobulin E (IgE) Antibodies | Baseline
Immunological Biomarkers | 4 months postpartum, 12 months postpartum
Medically-confirmed adverse events collected throughout the study period | 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei Liu, M.D., Principal Investigator — International Peace Maternity and Child Health Hospital of China Welfare Institution; Huiyong Yin, Ph.D., Principal Investigator — Chinese Academy of Sciences; Bryan Liu, Ph.D., Study Director — Mead Johnson & Company
Locations (1):
- International Peace Maternity and Child Health Hospital of China welfare Institute, Shanghai, Shanghai Municipality, China